CLINICAL TRIAL: NCT01083940
Title: Evaluating the Impact of Computerized Decision Support on Racial/Ethnic Disparities in Hypertension Outcomes
Brief Title: Impact of Computerized Decision Support on Racial/Ethnic Disparities in Hypertension Outcomes
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: LeRoi Hicks, MD, MPH, Brigham and Women's Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 66708
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reminders to providers (Experimental)
  Interventions: Other: Computerized reminders on hypertension intensification
- usual care (No Intervention)

INTERVENTIONS:
Other: Computerized reminders on hypertension intensification — Reminder generated to prompt providers to intensify therapy when patient's blood pressure remains uncontrolled
  Arms: Reminders to providers

SUMMARY:
In response to the Finding Answers: Disparities Research for Change call for proposals by the Robert Wood Johnson Foundation, we were funded to evaluate the effectiveness of a planned computerized decision support (CDS) intervention aimed at medical providers to overcome clinical inertia when treating blood pressure for hypertensive patients. Based on prior evaluation of the Brigham and Women's Hospital (BWH) adult primary care clinics, we hypothesize that racial and ethnic differences in blood pressure outcomes are largely attributable in differences in providers' aggressiveness in managing patients with hypertension based on patients' race and ethnicity. Within our network of 14 hospital and community-based Brigham and Women's Hospital adult primary care clinics, we aim to determine if the use of CDS to remind to medical providers of poorly controlled hypertensive patients to intensify their hypertension therapy will improve overall rates of blood pressure control and reduce the previously documented racial and ethnic disparities in blood pressure outcomes among our hypertensive patient population. Clinics will first be stratified by location (hospital-based versus community-based) and within each strata will be randomized to either have their providers receive CDS for hypertensive patients whose most recent blood pressure was uncontrolled or to usual care for hypertensive patients. More specifically, we will evaluate our planned intervention by utilizing an 18 month cluster-randomized controlled trial to examine the effectiveness the CDS for intensification of hypertension therapy in: improving levels of blood pressure control, improving provider adherence with recommended changes in drug therapy, and reducing racial/ethnic disparities in the processes of hypertension care and outcomes among our patients receiving primary care for a diagnosis of hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 20 years) with ICD-9 of hypertension with a minimum of 2 outpatient primary care visits in from 10/2008-10/2009 who receive care for hypertension in the outpatient practices at least once for hypertension from 10/2009-7/2001

Exclusion Criteria:

* Pregnancy, age < 20 years, fewer than two hypertension-related visits from 10/2008-10/2009

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3600 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Rate of blood pressure control at outcome between study arms | 10/1/2010-10/1/2011

SECONDARY OUTCOMES:
Rate of appropriate intensification of antihypertensive therapy | 10/2010-7/2011

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States